CLINICAL TRIAL: NCT04468581
Title: Characteristics of TraceTogether Users
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: 510d
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus
Keywords: Contact tracing; TraceTogether; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: We plan to recruit a representative sample of the Singapore population.
  Interventions: Behavioral: Use of mobile application

INTERVENTIONS:
Behavioral: Use of mobile application — Use of the TraceTogether mobile application during the COVID-19 period

SUMMARY:
In this protocol, we seek the understand the demographics of individuals who have used the TraceTogether mobile application. Little is known about the group of individuals who are more likely to utilise the application. Hence, this study hopes to: (1) Understand the demographics of Singaporeans who use and do not use TraceTogether, (2) Identify other behavioural habits of people who do use TraceTogether, (3) Determine if confidence in government would have any effect on TraceTogether usage

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years
* Has stayed in Singapore for at least 2 years

Exclusion Criteria:

* Below 21 years
* Has stayed in Singapore for less than 2 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative sample of the Singapore population
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Demographic information | Once during initial enrolment
  Age, gender, social economic status

CONTACTS AND LOCATIONS:
Locations (1):
- Yale NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the Institutional Review Board, data cannot be shared.

REFERENCES:
- [Derived] Saw YE, Tan EY, Liu JS, Liu JC. Predicting Public Uptake of Digital Contact Tracing During the COVID-19 Pandemic: Results From a Nationwide Survey in Singapore. J Med Internet Res. 2021 Feb 3;23(2):e24730. doi: 10.2196/24730. PMID 33465034